CLINICAL TRIAL: NCT02802995
Title: Safety And Efficacy Of Topical Platelet Rich Plasma And Thrombin Coagulum In The Treatment Of Recalcitrant Venous Stasis Ulcers
Brief Title: Safety And Efficacy Of Topical Platelet Rich Plasma And Thrombin Coagulum
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Resource issue
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Johnny Mahlangu, Professor, University of Witwatersrand, South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BDU005
Record Dates: First submitted 2016-05-17; First posted 2016-06-16 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2016-06

CONDITIONS: Stasis Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Subjects receiving the study drug which is PRP/thrombin mixture
  Interventions: Drug: PRP/thrombin mixture
- Control arm (No Intervention): Subjects receiving the standard of care for chronic venous wounds

INTERVENTIONS:
Drug: PRP/thrombin mixture — Mixture of platelet rich plasma and thrombin applied topically on the wound surface
  Other Names: thrombostim
  Arms: Treatment arm

SUMMARY:
The aim of this study is to

* To evaluate the safety and tolerability of Platelet Rich plasma(PRP)/Thrombin mixture in treating chronic venous ulcers
* To evaluate efficacy of PRP/Thrombin mixture in treating chronic venous ulcers

DETAILED DESCRIPTION:
Study rationale

In normal wound healing, platelets activate macrophages to produce endogenous platelet derived growth factor (PDGF) and other growth factors which are responsible for would healing. In chronic wounds, macrophage activation is suppressed which leads to an inappropriate growth factor response causing failure of positive autocrine feedback loop which normally controls the healing process. The regular application of exogenous PRP and Thrombin, to chronic wounds, restores the autocrine feedback loop of tissue repair which appears to accelerate the normal cascade of tissue repair

Objectives

* To evaluate the safety and tolerability of PRP/Thrombin mixture in treating chronic venous ulcers
* To evaluate efficacy of PRP/Thrombin mixture in treating chronic venous ulcers

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Age 18 years to 75 years.
* Both males and females.
* Ankle branchial index of 0.8 or above.

Exclusion Criteria:

* Diabetics will be excluded as the Ankle Branchial Index (ABI) result is considered an unreliable due the possible presence of arteriosclerotic plaques (lead pipe rigidity).
* Patients who have participated in experimental drug studies within 30 days of entering this study.
* receiving chemotherapy or radiotherapy for malignant diseases or any other indication
* Patients taking corticosteroids or other immunosuppressive medications
* Clinically malnourished patients or those with recent (last 4 weeks without treatment) serum albumin of less than 30g/l.
* Patients with current or past history of acute deep vein thrombosis.
* Patients with current signs and/or symptoms of cardiac, renal or hepatic failure. Renal failure defines as Creatinine
* Patients with signs and/or symptoms of peripheral neuropathy.
* Patients with signs and/or symptoms of ATROPHIE BLANCHE or other conditions associated with non-chronic venous insufficiency ulceration of the lower leg.
* Patients with signs and/or symptoms of immunocompromized sates or recent (last 4 weeks ) T cell subset (CD4) count of less than 200 cells / ml.
* Patients showing clinical signs and/or symptoms of anaemia or current or recent(last 4 weeks without treatment) haemoglobin level of less than 8g/dl

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Size of the wound treated with the PRP/thrombin mixture | 12 weeks
  Size of the wound will be measured at the end of the study
Number and type adverse events | 12 weeks
  Adverse events will reported at the start and throughout the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Mahlangu, MBBCH, MMed, Principal Investigator — Univeristy of the Witwatersrand
Locations (1):
- Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Callam MJ, Ruckley CV, Harper DR, Dale JJ. Chronic ulceration of the leg: extent of the problem and provision of care. Br Med J (Clin Res Ed). 1985 Jun 22;290(6485):1855-6. doi: 10.1136/bmj.290.6485.1855. PMID 3924283
- [Background] Dolynchuk K, Keast D, Campbell K, Houghton P, Orsted H, Sibbald G, Atkinson A. Best practices for the prevention and treatment of pressure ulcers. Ostomy Wound Manage. 2000 Nov;46(11):38-52; quiz 53-4. PMID 11889736
- [Background] Franz RC. Platelet concentrate-thrombin coagulum: a new biological dressing for the promotion of wound healing. S Afr Med J. 1987 Dec 5;72(11):810-1. No abstract available. PMID 3686285
- [Background] Franz RW, Shah KJ, Halaharvi D, Franz ET, Hartman JF, Wright ML. A 5-year review of management of lower extremity arterial injuries at an urban level I trauma center. J Vasc Surg. 2011 Jun;53(6):1604-10. doi: 10.1016/j.jvs.2011.01.052. Epub 2011 Apr 8. PMID 21477966
- [Background] Hammermeister KE, Johnson R, Marshall G, Grover FL. Continuous assessment and improvement in quality of care. A model from the Department of Veterans Affairs Cardiac Surgery. Ann Surg. 1994 Mar;219(3):281-90. doi: 10.1097/00000658-199403000-00008. PMID 8147609
- [Background] Hess CT. Pressure ulcer evidence-based treatment pathway integrated with evidence-based decisions: part 3. Adv Skin Wound Care. 2013 Sep;26(9):432. doi: 10.1097/01.ASW.0000434207.28117.5d. No abstract available. PMID 23958876
- [Background] Phillips LG, Mann R, Heggers JP, Linares HA, Robson MC. In vivo ovine flap model to evaluate surgical infection and tissue necrosis. J Surg Res. 1994 Jan;56(1):1-4. doi: 10.1006/jsre.1994.1001. PMID 8277759
- [Background] Pierce GF, Mustoe TA, Altrock BW, Deuel TF, Thomason A. Role of platelet-derived growth factor in wound healing. J Cell Biochem. 1991 Apr;45(4):319-26. doi: 10.1002/jcb.240450403. PMID 2045423
- [Background] Pierce GF, Brown D, Mustoe TA. Quantitative analysis of inflammatory cell influx, procollagen type I synthesis, and collagen cross-linking in incisional wounds: influence of PDGF-BB and TGF-beta 1 therapy. J Lab Clin Med. 1991 May;117(5):373-82. PMID 2019792
- [Background] Roe DF, Gibbins BL, Ladizinsky DA. Topical dissolved oxygen penetrates skin: model and method. J Surg Res. 2010 Mar;159(1):e29-36. doi: 10.1016/j.jss.2009.10.039. Epub 2009 Nov 21. PMID 20097370
- [Background] Steed DL, Ricotta JJ, Prendergast JJ, Kaplan RJ, Webster MW, McGill JB, Schwartz SL. Promotion and acceleration of diabetic ulcer healing by arginine-glycine-aspartic acid (RGD) peptide matrix. RGD Study Group. Diabetes Care. 1995 Jan;18(1):39-46. doi: 10.2337/diacare.18.1.39. PMID 7698046
- [Background] Wieman TJ, Smiell JM, Su Y. Efficacy and safety of a topical gel formulation of recombinant human platelet-derived growth factor-BB (becaplermin) in patients with chronic neuropathic diabetic ulcers. A phase III randomized placebo-controlled double-blind study. Diabetes Care. 1998 May;21(5):822-7. doi: 10.2337/diacare.21.5.822. PMID 9589248
- [Background] Wilkins RG, Unverdorben M. Wound cleaning and wound healing: a concise review. Adv Skin Wound Care. 2013 Apr;26(4):160-3. doi: 10.1097/01.ASW.0000428861.26671.41. PMID 23507692
- [Result] Atri SC, Misra J, Bisht D, Misra K. Use of homologous platelet factors in achieving total healing of recalcitrant skin ulcers. Surgery. 1990 Sep;108(3):508-12. PMID 2396195